CLINICAL TRIAL: NCT01196390
Title: A Phase III Trial Evaluating the Addition of Trastuzumab to Trimodality Treatment of HER2-Overexpressing Esophageal Adenocarcinoma
Brief Title: Radiation Therapy, Paclitaxel, and Carboplatin With or Without Trastuzumab in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02601; NCI-2011-02601 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000683717; RTOG-1010; RTOG-1010 (Other: NRG Oncology); RTOG-1010 (Other: CTEP); U10CA180830 (NIH); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Stage IB Esophageal Cancer AJCC v7; Stage IIA Esophageal Cancer AJCC v7; Stage IIB Esophageal Cancer AJCC v7; Stage IIIA Esophageal Cancer AJCC v7; Stage IIIB Esophageal Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; Radiotherapy; Radiation; Trastuzumab; CT-P6; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (radiotherapy, chemotherapy, trastuzumab) (Experimental): Patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Patients also receive trastuzumab IV over 30-90 minutes on days 1, 8, 15, 22, 29, 36, and 57 and paclitaxel intravenously IV over 60 minutes and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Beginning 21-56 days after surgery, patients receive trastuzumab IV over 30-90 minutes. Treatment repeats every 21 days for 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab
- Arm II (radiotherapy and chemotherapy) (Experimental): Patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Patients also receive paclitaxel IV over 60 minutes and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; Ogivri; Ontruzant; PF-05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
  Arms: Arm I (radiotherapy, chemotherapy, trastuzumab)

SUMMARY:
This randomized phase III trial studies how well radiation therapy, paclitaxel, and carboplatin with or without trastuzumab work in treating patients with esophageal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as trastuzumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving radiation therapy and combination chemotherapy together with or without trastuzumab is more effective in treating esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To determine if trastuzumab increases disease-free survival when combined with trimodality treatment (radiation plus chemotherapy followed by surgery) for patients with human epidermal growth factor receptor 2 (HER2)-overexpressing esophageal adenocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate if the addition of trastuzumab to trimodality treatment increases the pathologic complete response rate and overall survival for patients with HER2-overexpressing esophageal adenocarcinoma.

II. To develop a tissue bank of tumor tissue from patients with non-metastatic esophageal adenocarcinoma.

III. To determine molecular correlates of complete pathologic response, disease-free survival, and overall survival for patients with HER2-overexpressing esophageal adenocarcinoma treated with neoadjuvant and maintenance trastuzumab.

IV. To evaluate predictors of cardiotoxicity in patients with esophageal cancer treated with trastuzumab and chemoradiation.

V. To evaluate adverse events associated with the addition of trastuzumab to trimodality treatment for patients with non-metastatic esophageal adenocarcinoma.

PATIENT-REPORTED QUALITY OF LIFE OBJECTIVES:

I. To determine if the addition of trastuzumab to trimodality treatment improves the patient-reported Functional Assessment of Cancer Therapy for Esophageal Cancer (FACT-E) Esophageal Cancer Subscale (ECS) score.

II. To determine if an improvement in the FACT-E ECS score at 6-8 weeks post completion of neoadjuvant chemoradiation correlates with pathologic complete response.

III. To determine if pathologic complete response correlates with the FACT-E ECS score at 1 year and/or 2 years from the start of chemoradiation.

IV. To determine if the addition of trastuzumab to trimodality treatment improves the Swallow Index and Eating Index Subscale scores of the FACT-E.

V. To determine if the addition of trastuzumab to paclitaxel, carboplatin, and radiation impacts quality-adjusted survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Patients also receive trastuzumab intravenously (IV) over 30-90 minutes on days 1, 8, 15, 22, 29, 36, and 57 and paclitaxel IV over 60 minutes and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36. Beginning 21-56 days after surgery, patients receive trastuzumab IV over 30-90 minutes. Treatment repeats every 21 days for 13 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo radiotherapy once daily 5 days a week for 5.5 weeks. Patients also receive paclitaxel IV over 60 minutes and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36.

Within 5-8 weeks after completion of radiotherapy, all patients undergo surgery.

After completion of study therapy, patients are followed up every 4 months for 2 years and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed primary adenocarcinoma of the esophagus that involves the mid (up to 25 cm), distal, or esophagogastric junction; the cancer may involve the stomach up to 5 cm
* Endoscopy with biopsy
* PRIOR TO STEP 1 REGISTRATION BUT WITHIN 56 DAYS PRIOR TO STEP 2 REGISTRATION
* Intent to submit tissue for central HER2 testing
* Stage T1N1-2, T2-3N0-2, according to the American Joint Committee on Cancer (AJCC) 7th edition staging, based on the following minimum diagnostic work-up:

  * Chest/abdominal/pelvic computed tomography (CT) or whole-body positron emission tomography (PET)/CT (NOTE: if CT is performed at this time point, whole-body PET/CT will be required prior to step 2 registration; PET/CT of skull base to mid-thigh is acceptable) (NOTE: if adenopathy is noted on CT or whole-body PET/CT scan, an endoscopic ultrasound is not required prior to STEP 2 registration as long as adequate tissue has been obtained for central HER2 testing)
  * Patients may have regional adenopathy including para-esophageal, gastric, gastrohepatic and celiac nodes; if celiac adenopathy is present, it must be =< 2 cm
  * Patients with tumors at the level of the carina or above must undergo bronchoscopy to exclude fistula
* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 8.0 g/dL (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dL is acceptable)
* Creatinine =< 2 times upper limit of normal
* Bilirubin =< 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) =< 3.0 times upper limit of normal
* For women of childbearing potential, a negative serum or urine pregnancy test
* Patients must sign a study-specific informed consent prior to study entry
* CONDITIONS FOR PATIENT ELIGIBILITY PRIOR TO STEP 2 REGISTRATION (HER2-POSITIVE PATIENTS ONLY)
* HER2 expressing adenocarcinoma of the esophagus centrally
* Surgical consultation to confirm that patient will be able to undergo curative resection after completion of chemoradiation within 56 days prior to step 2 registration
* Radiation oncology consultation to confirm that disease can be encompassed in a radiotherapy field within 56 days prior to step 2 registration
* Consultation with a medical oncologist within 56 days prior to step 2 registration
* Stage T1N1-2, T2-3N0-2, according to the AJCC 7th edition staging, based upon the following minimum diagnostic work-up:

  * History/physical examination, with documentation of the patient's weight, within 14 days prior to step 2 registration
  * Whole-body PET/CT scan within 56 days prior to step 2 registration (if only CT performed prior to step 1 registration)
  * Endoscopic ultrasound within 56 days prior to step 2 registration, unless the patient is found to have adenopathy per CT or whole-body PET/CT scan
  * Electrocardiogram (EKG) within 56 days prior to step 2 registration
  * Serum creatinine =< 2 x the upper limit or normal within 14 days prior to step 2 registration
* Zubrod performance status 0-2 within 14 days prior to step 2 registration
* For women of childbearing potential, a negative serum pregnancy test within 14 days prior to step 2 registration
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal by cardiac echocardiogram (echo) or multi gated acquisition (MUGA) scan within 56 days prior to step 2 registration
* Women of childbearing potential and sexually active male participants must agree to practice adequate contraception while on study and for at least 60 days following the last dose of chemotherapy or trastuzumab

Exclusion Criteria:

* Patients with cervical esophageal carcinoma
* Patients with T1N0 disease, T4 disease, and proximal esophageal cancers (15-24 cm)
* Prior systemic chemotherapy for esophageal cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiation therapy for esophageal cancer or prior chest radiotherapy
* Prior anthracycline or taxane
* Evidence of tracheoesophageal fistula or invasion into the trachea or major bronchi
* Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 2 years (e.g., carcinoma in situ of the breast, oral cavity, or cervix are permissible)
* Medical contraindications to esophagectomy
* Prior therapy with any agent targeting the HER2 pathway or human epidermal growth factor receptor 1 (HER1) (epidermal growth factor receptor [EGFR]) pathway
* Prior therapy with trastuzumab
* Prior allergic reaction to the study drugs involved in this protocol or to a monoclonal antibody
* Previous history of congestive heart failure
* Severe, active comorbidity, defined as follows:

  * Unstable angina in the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; protocol-specific requirements may also exclude immunocompromised patients
* Pregnant or nursing women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2011-02-14 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard P Safran, Principal Investigator — NRG Oncology
Locations (634):
- United States (634):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Concord Hospital, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - American College of Radiology Imaging Network, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiation Oncology Associates Incorporated, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Safran HP, Winter K, Ilson DH, Wigle D, DiPetrillo T, Haddock MG, Hong TS, Leichman LP, Rajdev L, Resnick M, Kachnic LA, Seaward S, Mamon H, Diaz Pardo DA, Anderson CM, Shen X, Sharma AK, Katz AW, Salo J, Leonard KL, Moughan J, Crane CH. Trastuzumab with trimodality treatment for oesophageal adenocarcinoma with HER2 overexpression (NRG Oncology/RTOG 1010): a multicentre, randomised, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):259-269. doi: 10.1016/S1470-2045(21)00718-X. Epub 2022 Jan 14. PMID 35038433
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After registration, sites were required to submit participant tumor tissue for central human epidermal growth factor receptor 2 (HER2) testing. Only HER2-positive participants continued to randomization. In total, 571 participants were registered and 203 were randomized.
Groups:
- Chemoradiation and Trastuzumab: Radiation therapy with concurrent trastuzumab, paclitaxel, and carboplatin followed by surgery followed by maintenance trastuzumab
- Chemoradiation: Radiation therapy with concurrent paclitaxel and carboplatin followed by surgery
Period: Overall Study
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Started | 102 | 101
Eligible | 98 | 96
Eligible and Started Study Treatment | 95 | 96
Eligible and Had Surgery | 82 | 78
Eligible and Consented to Quality of Life Component | 88 | 83
Completed (Participants contributing data to results are considered to have completed the study) | 98 | 96
Not Completed | 4 | 5
Not completed — Protocol Violation | 4 | 5

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Customized [Count of Participants; unit: Participants]
  ≤ 39 years | 0 | 5 | 5
  40-49 years | 6 | 7 | 13
  50-59 years | 30 | 21 | 51
  60-69 years | 40 | 31 | 71
  70-79 years | 20 | 29 | 49
  ≥ 80 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 85 | 79 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 96 | 89 | 185
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 94 | 92 | 186
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 62 | 62 | 124
    1 | 34 | 31 | 65
    2 | 2 | 3 | 5
T stage, clinical [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 1 | 4 | 5
    T2 | 18 | 17 | 35
    T3 | 79 | 75 | 154
N stage, clinical [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes.
  Participants
    N0 | 27 | 29 | 56
    N1 | 55 | 48 | 103
    N2 | 16 | 19 | 35
Presence of Adenopathy [Count of Participants; unit: Participants]
  No | 38 | 38 | 76
  Yes adenopathy, but celiac absent | 48 | 48 | 96
  Yes adenopathy and celiac present ≤ 2 cm | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: A disease event is defined as local/regional persistence or recurrence of the cancer under study, distant metastases, a new second primary cancer, or death due to any cause. Participants undergoing surgery who had an R2 resection and participants not undergoing surgery who had a positive endoscopic biopsy or no biopsy at all were considered to have local persistence of disease. Disease-free survival time is defined as time from randomization to the date of first disease event or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. Analysis was to occur after 162 events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 8.0 years.
Population: Eligible randomized participants
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Chemoradiation and Trastuzumab (Arm 1): Radiation therapy with concurrent trastuzumab, paclitaxel, and carboplatin followed by surgery followed by maintenance trastuzumab
- Chemoradiation (Arm 2): Radiation therapy with concurrent paclitaxel and carboplatin followed by surgery
Arm/Group | Chemoradiation and Trastuzumab (Arm 1) | Chemoradiation (Arm 2)
Number analyzed (Participants) | 98 | 96
months | 19.6 [13.5 to 26.2] | 14.2 [10.5 to 23.0]
Statistical Analysis 1: Comparison: Chemoradiation and Trastuzumab (Arm 1) vs Chemoradiation (Arm 2); Assuming a median DFS time of 15 months (Arm 2), hypothesized increase in DFS corresponding to median DFS time of 25 months (Arm 1). Assuming an exponential distribution and constant hazards, 183 HER2-positive participants accrued over 5 years and followed for 3 years would result in 162 disease-free survival events and provide 90% statistical power to detect this difference with a 2-sided α of 0.05 and 2 interim analyses. See Limitations and Caveats section; Test type: Superiority; p = 0.85, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.69 to 1.36] — Reference level = Chemoradiation arm

2. Secondary Outcome: Percentage of Participants With Pathologic Complete Response at Surgery
Description: Pathologic Complete Response (pCR) is evaluated after surgery and is based on the pathology review of the submitted surgical specimen. Pathologic Complete Response occurs if the pathologist determines that the resected esophageal specimen, accompanying lymph nodes, and surgical margins are all free of tumor.
Time Frame: At the time of surgery, 5-8 weeks after completion of radiation therapy.
Population: Eligible participants who had surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 82 | 78
percentage of participants | 27 [18 to 38] | 29 [20 to 41]
Statistical Analysis 1: Comparison: Chemoradiation and Trastuzumab vs Chemoradiation; Test type: Superiority; p = 0.71, Chi-squared; Two-sided significance level = 0.05

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. Analysis occurred after 109 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 8 years.
Population: Eligible randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 98 | 96
months | 38.5 [26.2 to 70.4] | 38.9 [29.0 to 64.5]
Statistical Analysis 1: Comparison: Chemoradiation and Trastuzumab vs Chemoradiation; Test type: Superiority; p = 0.95, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.69 to 1.47] — Reference level = Chemoradiation arm

4. Secondary Outcome: Frequency of Highest Grade Adverse Event Per Participant
Description: Common Terminology Criteria for Adverse Events (version 4.0 before 4-1-2018; then version 5.0) grades adverse event severity from 1=mild to 5=death. Summary data provided is in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 8 years.
Population: Eligible participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 95 | 96
Participants
  All Adverse Events: Grade 1 | 0 | 0
  All Adverse Events: Grade 2 | 14 | 12
  All Adverse Events: Grade 3 | 49 | 56
  All Adverse Events: Grade 4 | 27 | 25
  All Adverse Events: Grade 5 | 5 | 3
  Reported as Definitely, Probably, or Possibly Related to Protocol Treatment: Grade 1 | 2 | 0
  Reported as Definitely, Probably, or Possibly Related to Protocol Treatment: Grade 2 | 27 | 20
  Reported as Definitely, Probably, or Possibly Related to Protocol Treatment: Grade 3 | 41 | 52
  Reported as Definitely, Probably, or Possibly Related to Protocol Treatment: Grade 4 | 20 | 21
  Reported as Definitely, Probably, or Possibly Related to Protocol Treatment: Grade 5 | 5 | 3

5. Secondary Outcome: Percentage of Patients With Improvement in the Functional Assessment of Cancer Therapy - Esophagus (FACT-E) Esophageal Cancer Subscale (ECS) Subscale After Treatment
Description: The ECS is a 17-item self-report instrument designed to measure multidimensional quality of life in patients with esophagus cancer with a total score ranging from 0-68. It is to be administered with the Functional Assessment of Cancer Therapy - General (FACT-G). A higher score indicates better QOL. Improvement is defined as an increase from the baseline score of at least 5 points.
Time Frame: Baseline, 6-8 weeks after end of radiation therapy (approximately 11.5-13.5 weeks from treatment start), 1 and 2 years from treatment start
Population: Eligible participants who consented to quality of life evaluation and who had baseline and time point data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 88 | 83
percentage of participants
  6-8 weeks from end of treatment: number analyzed (Participants) | 48 | 56
  6-8 weeks from end of treatment | 46 [33 to 60] | 38 [26 to 51]
  1 year from start of treatment: number analyzed (Participants) | 44 | 36
  1 year from start of treatment | 39 [26 to 53] | 42 [27 to 58]
  2 years from start of treatment: number analyzed (Participants) | 22 | 30
  2 years from start of treatment | 41 [23 to 61] | 27 [14 to 45]
Statistical Analysis 1: Comparison: Chemoradiation and Trastuzumab vs Chemoradiation; 6-8 weeks; Test type: Superiority; p = 0.39, Chi-squared — One-side significance level = 0.05
Statistical Analysis 2: Comparison: Chemoradiation and Trastuzumab vs Chemoradiation; 1 year; Test type: Superiority; p = 0.78, Chi-squared — One-side significance level = 0.05
Statistical Analysis 3: Comparison: Chemoradiation and Trastuzumab vs Chemoradiation; 2 years; Test type: Superiority; p = 0.28, Chi-squared — One-side significance level = 0.05

6. Secondary Outcome: Quality-adjusted Survival
Time Frame: From randomization to last follow-up. Maximum follow-up at time of primary outcome measure analysis was 8 years.
Population: The protocol states that this outcome measure will be analyzed only if primary outcome results are positive, i.e. support the primary hypothesis of this study. Therefore no participants were analyzed for this outcome measure.
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Molecular Correlates of Efficacy
Time Frame: From randomization to last follow-up. Maximum follow-up at time of primary outcome measure analysis was 8 years.
Population: The protocol did not provide sufficient detail to meet current National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed, and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Any Cardiac Adverse Events Regardless of Attribution
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event (AE) severity from 1=mild to 5=death. Logistic regression was used to evaluate treatment arm, clinical tumor stage (T stage), Zubrod Performance Status, gender, presence of adenopathy, and age as possible predictors of cardiac adverse events. Results of the final model are reported in the statistical analysis section. Summary adverse event data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 8 years.
Population: Eligible participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiation and Trastuzumab (Arm 1) | Chemoradiation (Arm 2)
Number analyzed (Participants) | 95 | 96
Participants | 30 | 24
Statistical Analysis 1: Comparison: Chemoradiation and Trastuzumab (Arm 1) vs Chemoradiation (Arm 2); Logistic regression was used to model the association of treatment arm (Arm 1 vs. 2 [reference level(RL)]), T stage (T3 vs.T1,T2 [RL]), Zubrod (1,2 vs. 0 [RL]), gender (male vs. female [RL]), presence of adenopathy (yes vs. no [RL]), and age (≥ 60 vs. <60 [RL]) with the occurrence of any cardiac AE, using backwards step-wise model selection requiring p≤0.05 for a covariate to remain in the model. Final model covariates are reported. Age is reported here. No other covariates reported; Test type: Superiority; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.13 to 4.86]

ADVERSE EVENTS:
Time Frame: Day 8, 15, 22, 29, and 36 and completion (day 57) of concurrent chemoradiation, before surgery (5-8 weeks after last radiation treatment), every 4 mos from the end of surgery for 2 years, then annually until study completion. Maximum follow-up at time of analysis was 8.0 years.
Arm/Group | Chemoradiation and Trastuzumab | Chemoradiation
All-Cause Mortality (participants affected / at risk) | 53/95 | 55/96
Serious Adverse Events (participants affected / at risk) | 51/95 | 34/96
Other Adverse Events (participants affected / at risk) | 95/95 | 96/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation and Trastuzumab (N=95) | Chemoradiation (N=96)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 4
Esophageal fistula (Gastrointestinal disorders) | 2 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Esophageal perforation (Gastrointestinal disorders) | 1 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 3 | 3
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 6
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Fever (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Sudden death NOS (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 3 | 3
Pleural infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 2
Stoma site infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 3 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 4
Neutrophil count decreased (Investigations) | 4 | 3
Platelet count decreased (Investigations) | 1 | 1
Urine output decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 3
White blood cell decreased (Investigations) | 4 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 2
Thromboembolic event (Vascular disorders) | 3 | 2
Visceral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation and Trastuzumab (N=95) | Chemoradiation (N=96)
Anemia (Blood and lymphatic system disorders) | 61 | 57
Atrial fibrillation (Cardiac disorders) | 5 | 3
Cardiac disorders - Other, specify (Cardiac disorders) | 3 | 5
Sinus tachycardia (Cardiac disorders) | 6 | 9
Abdominal pain (Gastrointestinal disorders) | 28 | 31
Bloating (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 38 | 45
Diarrhea (Gastrointestinal disorders) | 42 | 36
Dry mouth (Gastrointestinal disorders) | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 27 | 16
Dysphagia (Gastrointestinal disorders) | 57 | 50
Esophageal pain (Gastrointestinal disorders) | 13 | 13
Esophageal stenosis (Gastrointestinal disorders) | 8 | 4
Esophagitis (Gastrointestinal disorders) | 52 | 41
Gastritis (Gastrointestinal disorders) | 7 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 19 | 11
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 13 | 11
Gastrointestinal pain (Gastrointestinal disorders) | 6 | 1
Mucositis oral (Gastrointestinal disorders) | 13 | 14
Nausea (Gastrointestinal disorders) | 66 | 69
Vomiting (Gastrointestinal disorders) | 32 | 33
Chills (General disorders) | 12 | 11
Edema limbs (General disorders) | 13 | 7
Fatigue (General disorders) | 78 | 71
Fever (General disorders) | 12 | 11
General disorders and administration site conditions - Other, specify (General disorders) | 7 | 2
Infusion related reaction (General disorders) | 8 | 6
Non-cardiac chest pain (General disorders) | 8 | 7
Pain (General disorders) | 22 | 18
Lung infection (Infections and infestations) | 4 | 6
Skin infection (Infections and infestations) | 3 | 5
Upper respiratory infection (Infections and infestations) | 8 | 4
Urinary tract infection (Infections and infestations) | 5 | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 | 10
Alanine aminotransferase increased (Investigations) | 10 | 9
Alkaline phosphatase increased (Investigations) | 15 | 8
Aspartate aminotransferase increased (Investigations) | 16 | 9
Blood bilirubin increased (Investigations) | 5 | 8
Creatinine increased (Investigations) | 3 | 5
Lymphocyte count decreased (Investigations) | 40 | 37
Neutrophil count decreased (Investigations) | 47 | 50
Platelet count decreased (Investigations) | 58 | 64
Weight loss (Investigations) | 45 | 45
White blood cell decreased (Investigations) | 78 | 81
Anorexia (Metabolism and nutrition disorders) | 41 | 46
Dehydration (Metabolism and nutrition disorders) | 24 | 22
Hyperglycemia (Metabolism and nutrition disorders) | 37 | 31
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 7
Hypernatremia (Metabolism and nutrition disorders) | 6 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 20 | 19
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 15 | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 11
Hyponatremia (Metabolism and nutrition disorders) | 31 | 24
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 18
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Dizziness (Nervous system disorders) | 20 | 15
Dysgeusia (Nervous system disorders) | 13 | 19
Headache (Nervous system disorders) | 10 | 12
Nervous system disorders - Other, specify (Nervous system disorders) | 6 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 18
Anxiety (Psychiatric disorders) | 18 | 12
Depression (Psychiatric disorders) | 10 | 10
Insomnia (Psychiatric disorders) | 18 | 23
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 24
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 14
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 13 | 2
Hypertension (Vascular disorders) | 8 | 15
Hypotension (Vascular disorders) | 13 | 14
Thromboembolic event (Vascular disorders) | 2 | 6

LIMITATIONS AND CAVEATS:
Due to a considerable decrease in the overall rate of new disease-free survival events, the NRG Data Monitoring Committee (DMC) determined that the study would not reach the required 162 events in a reasonable amount of time. With power from the observed number of events calculated to be greater than 80%, the DMC recommended releasing the results for reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT01196390/Prot_SAP_000.pdf